CLINICAL TRIAL: NCT00954005
Title: Multicentric Phase I/II Study for the Efficacy of a Combination of Rituximab, Gemcitabine and Oxaliplatin in Relapsed/Refractory Indolent Lymphoma
Brief Title: Study With Rituximab-Gemcitabine/Oxaliplatin in Relapsed Indolent Lymphoma
Acronym: R-GO
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Predefined termination criterion of > 10 patients without CR or PR was matched.
Sponsor: German Low Grade Lymphoma Study Group (Other)
Responsible Party: Principal Investigator, Martin Hoffmann, Dr. Martin Hoffmann, Klinikum Ludwigshafen, German Low Grade Lymphoma Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Indolent Lymphoma
Keywords: relapsed indolent lymphoma; gemcitabine; oxaliplatin; rituximab
MeSH Terms: interventions — Therapeutics; Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab, Gemcitabine and Oxaliplatin (Experimental): Drug: Rituximab on day 0 or 1 of each 28-day cycle Drug: Gemcitabine on day 1 and 15 of each 28-day cycle Drug: Oxaliplatin on day 1 and 15 (in phase 1 dose escalation of Oxaliplatin in steps of 10 mg/m²) of each 28-day cycle
  Interventions: Drug: Therapy with Rituximab, Gemcitabine and Oxaliplatin

INTERVENTIONS:
Drug: Therapy with Rituximab, Gemcitabine and Oxaliplatin — Rituximab 375 mg/m² day 0 or 1, Gemcitabine 1.000 mg/m² in 30 Min. day 1 and 15, Oxaliplatin 70 mg/m² in 120 Min. day 1 and 15 (in phase 1 dose escalation of Oxaliplatin in steps of 10 mg/m²), repetition at day 29 for 4 cycles
  Other Names: Rituximab = Mabthera, Rituxan; Gemcitabine = Gemzar; Oxaliplatin = Eloxatin

SUMMARY:
The purpose of the phase I part is to determine the tolerability, the initial safety profile and maximum tolerated dose of oxaliplatin in combination with gemcitabine for indolent lymphoma. In the phase II part the investigators want to estimate the activity of gemcitabine and oxaliplatin in combination with rituximab for patients with relapsed/refractory indolent lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Need for therapy in patients with relapsed/refractory patients
* Histological proven diagnosis of an indolent B-cell lymphoma according to the World Health Organization (WHO) classification belonging to one of the following entities:

  * follicular lymphoma
  * mantle cell lymphoma
  * lymphoplasmacytic lymphoma
  * nodal or splenic marginal zone lymphoma
  * measurable disease
  * lymphoma specific therapy in the last four weeks
  * WHO performance grade 0, 1 or 2

Exclusion Criteria

* Patients suitable for high dose therapy
* Transformation in high grade lymphoma
* Leukocytes < 1,5/nl or platelets < 100/nl (except due to lymphoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-01; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Overall Remission Rate | end of therapy

SECONDARY OUTCOMES:
Progression Free Survival | 5 years
Median Overall Survival | 5 years
Toxicity | 5 years
  Number of Participants With Treatment-Related Adverse Events as Assessed by WHO Toxicity Grading Scale

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hoffmann, Dr., Principal Investigator — German Low Grade Lymphoma Study Group
Locations (1):
- Klinikum Ludwigshafen, Ludwigshafen, Germany

REFERENCES:
- [Derived] Scheubeck G, Hoffmann M, Jurinovic V, Fischer L, Unterhalt M, Schmidt C, Bock HP, Duhrsen U, Kaesberger J, Kremers S, Lindemann HW, Mantovani L, Hiddemann W, Hoster E, Dreyling M; German Lymphoma Alliance (GLA). Rituximab, gemcitabine and oxaliplatin in relapsed or refractory indolent and mantle cell lymphoma: results of a multicenter phase I/II-study of the German Low Grade Lymphoma Study Group. Ann Hematol. 2024 Jul;103(7):2373-2380. doi: 10.1007/s00277-024-05689-w. Epub 2024 Mar 9. PMID 38459156